CLINICAL TRIAL: NCT06424938
Title: The Effect of Epidural Analgesia and Erector Spinae Plane Block on Intraoperative and Early Postoperative Outcomes in Open Gynecological Oncological Surgeries: a Prospective Randomized Study
Brief Title: Postoperative Analgesia in Major Gynecological Cancer Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duygu Akyol (Other Government)
Responsible Party: Sponsor-Investigator, Duygu Akyol, M.D, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Organization: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-597
Record Dates: First submitted 2024-05-14; First posted 2024-05-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-06

CONDITIONS: Analgesia; Analgesia, Epidural; ERAS
Keywords: postoperative analgesia; periferic nerve block; neuraxial block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: This study was designed as a prospective randomized study. Patients with ASA II-III between the ages of 30 and 70 who will undergo major gynecological cancer surgery will be included in the study. They will be randomized into 2 groups: the group in which epidural block is applied for postoperative analgesia (Group Epidural) and the group in which erector spinae plane block is applied (Group ESP).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group in which epidural block (Experimental): The group in which epidural block is applied for postoperative analgesia (Group Epidural)
  Interventions: Procedure: Patients who underwent epidural block; Procedure: Patients who underwent erector spina plane block
- The group in which erector spinae plane block (Experimental): The group in which erector spinae plane block is applied (Group ESP)
  Interventions: Procedure: Patients who underwent epidural block; Procedure: Patients who underwent erector spina plane block

INTERVENTIONS:
Procedure: Patients who underwent epidural block — The researchers administered an epidural block to prevent post-operative pain to the epidural block group undergoing midline incision surgery for major gynecologic cancer.
Procedure: Patients who underwent erector spina plane block — Researchers applied a erector spina plane block to prevent postoperative pain to the erector spina plane block group undergoing midline incision surgery for major gynecological cancer.

SUMMARY:
The aim of this study is to compare the effectiveness of epidural block or erector spinae plane block applied for postoperative analgesia in gynecological cancer surgeries.

The main question(s) it aims to answer are:

[Is erector spinae plane block as effective as epidural block in postoperative analgesia?] The study was designed as a prospective randomized study. Researchers evaluated the effects of epidural block or erector spinae plane block applied for postoperative analgesia on pain scores, postoperative opioid use, and mobilization in patients undergoing gynecological cancer surgery.

DETAILED DESCRIPTION:
Our study was designed as a prospective randomized study. The investigators evaluated the analgesia methods used in patients undergoing surgery for gynecologic cancer between May 2024 and December 2024. The investigators evaluated the effect of epidural block or erector spina plan block on postoperative analgesia, opioid use and mobilization.

Group 1: Epidural block group Group 2: Group with erector spina plan block

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo open abdominal surgery
* Patients with ASAII-III
* Those between the ages of 30-70
* Patients who are fully oriented and able to cooperate

Exclusion Criteria:

* Patients with ASAIV-V
* Presence of active infection in the area where the block will be applied
* Patients younger than 30 years old
* Patients with BMI > 40
* Patients who are allergic to bupivacaine
* Chronic analgesic use

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
postoperative numerical rating scale | postoperatvely 24 hours
  The primary purpose of this study is to compare NRS values at 0, 6, 12 and 24 hours in the first 24 hours postoperatively. Numeric rating scale was used to assess postoperative pain For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable.

SECONDARY OUTCOMES:
Intraoperative amount of remifentanyl | intraoperative process
  The secondary aim of this study is to compare the amount of intraoperative remifentanyl

OTHER OUTCOMES:
postoperative mobilization time | postoperatvely 24 hours
  The other purpose of this study is the first postoperative mobilization process

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson G, Fotopoulou C, Taylor J, Glaser G, Bakkum-Gamez J, Meyer LA, Stone R, Mena G, Elias KM, Altman AD, Bisch SP, Ramirez PT, Dowdy SC. Enhanced recovery after surgery (ERAS(R)) society guidelines for gynecologic oncology: Addressing implementation challenges - 2023 update. Gynecol Oncol. 2023 Jun;173:58-67. doi: 10.1016/j.ygyno.2023.04.009. Epub 2023 Apr 21. PMID 37086524
- [Background] Bisch SP, Jago CA, Kalogera E, Ganshorn H, Meyer LA, Ramirez PT, Dowdy SC, Nelson G. Outcomes of enhanced recovery after surgery (ERAS) in gynecologic oncology - A systematic review and meta-analysis. Gynecol Oncol. 2021 Apr;161(1):46-55. doi: 10.1016/j.ygyno.2020.12.035. Epub 2020 Dec 30. PMID 33388155
- [Background] Courtney-Brooks M, Tanner Kurtz KC, Pelkofski EB, Nakayama J, Duska LR. Continuous epidural infusion anesthesia and analgesia in gynecologic oncology patients: less pain, more gain? Gynecol Oncol. 2015 Jan;136(1):77-81. doi: 10.1016/j.ygyno.2014.10.015. Epub 2014 Oct 23. PMID 25449564
- [Background] Chen LM, Weinberg VK, Chen C, Powell CB, Chen LL, Chan JK, Burkhardt DH 3rd. Perioperative outcomes comparing patient controlled epidural versus intravenous analgesia in gynecologic oncology surgery. Gynecol Oncol. 2009 Dec;115(3):357-61. doi: 10.1016/j.ygyno.2009.08.015. Epub 2009 Sep 23. PMID 19783285
- [Background] Ferguson SE, Malhotra T, Seshan VE, Levine DA, Sonoda Y, Chi DS, Barakat RR, Abu-Rustum NR. A prospective randomized trial comparing patient-controlled epidural analgesia to patient-controlled intravenous analgesia on postoperative pain control and recovery after major open gynecologic cancer surgery. Gynecol Oncol. 2009 Jul;114(1):111-6. doi: 10.1016/j.ygyno.2009.03.014. Epub 2009 Apr 23. PMID 19395071
- [Background] Lin C, Gill R, Kumar K. [Bilateral lower thoracic erector spinae plane block in open abdominal gynecologic oncology surgery: a cases series]. Braz J Anesthesiol. 2019 Sep-Oct;69(5):517-520. doi: 10.1016/j.bjan.2019.03.011. Epub 2019 Oct 19. PMID 31635757